CLINICAL TRIAL: NCT06524063
Title: Phase I Clinical Study of Targeted Survivin DC Cell Injection for the Treatment of Newly Diagnosed Primary Glioblastoma Multiforme (GBM)
Brief Title: Targeted Survivin DC Cell Injection for the Treatment of GBM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tricision Biotherapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QCS-gc-001; CTR20240438 (Other: NMPA)
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivin-loaded dendritic cell injection (Experimental): Patients will undergo a combined treatment of radiotherapy and temozolomide (TMZ) for a duration of 6 weeks, with concurrent chemotherapy. After completing this phase, there will be a 4-week interval (28 days) before entering multiple cycles of adjuvant TMZ chemotherapy. Each cycle will last 28 days, involving daily oral administration of temozolomide at a dose of 150-200mg/m2 for 5 consecutive days, followed by a 23-day drug-free period. This entire cycle will be repeated every 28 days. Nine days after completing the standard 6-week concurrent chemoradiotherapy, targeted Survivin DC cell injections will be administered. The injections will be given on days 0, 14, and 28. The administration will involve both intradermal (ID) and intravenous (IV) routes.
  Interventions: Drug: Survivin-loaded dendritic cell injection

INTERVENTIONS:
Drug: Survivin-loaded dendritic cell injection — The injections will be given on days 0, 14, and 28. The administration will involve both intradermal (ID) and intravenous (IV) routes.
  Other Names: Targeted Survivin DC cell therapy

SUMMARY:
Primary Objective: To evaluate the safety and tolerability of targeted Survivin DC cell injection for postoperative treatment of newly diagnosed primary glioblastoma multiforme. Secondary Objectives: Utilize progression-free survival (PFS) and overall survival (OS) to preliminarily assess the effectiveness of targeted Survivin DC cell injection for postoperative treatment of newly diagnosed primary glioblastoma multiforme in China. Evaluate the immunological effects of targeted Survivin DC cell injection. Explore the impact of targeted Survivin DC cell injection on human DC cell activity and in vivo processes.

Patients will undergo a combined treatment of radiotherapy and temozolomide (TMZ) for a duration of 6 weeks, with concurrent chemotherapy. After completing this phase, there will be a 4-week interval (28 days) before entering multiple cycles of adjuvant TMZ chemotherapy. Each cycle will last 28 days, involving daily oral administration of temozolomide at a dose of 150-200mg/m2 for 5 consecutive days, followed by a 23-day drug-free period. This entire cycle will be repeated every 28 days. Nine days after completing the standard 6-week concurrent chemoradiotherapy, targeted Survivin DC cell injections will be administered. The injections will be given on days 0, 14, and 28. The administration will involve both intradermal (ID) and intravenous (IV) routes. Four hours before the administration, the injection sites will be pre-treated with lidocaine cream. The injection procedures will be conducted sequentially, starting with ID injection. After completing the ID injection, a 30-minute observation will be conducted. If no adverse reactions are observed, IV infusion will be initiated. Both IV infusion and ID injection will be performed on the same side. Intradermal Injection: Draw 1ml of cell suspension with a 1ml syringe, and the remaining cell product will be stored at 2-8℃. Administer the drug immediately after preparation. Intravenous Infusion: Before administration, infuse 20ml of normal saline through IV.Extract 25ml of normal saline, dilute the remaining cell product (5ml), and administer it through IV infusion. Control the room temperature during infusion and complete it within 30 minutes. After administration, inject 50ml of normal saline into the cell bag to ensure all cell products are returned to the patient's body.

DETAILED DESCRIPTION:
The trial was designed as an open-label, dose-escalation trial. This study is divided into two phases: a dose escalation phase and an expansion cohort phase.

Dose escalation phase: This project is for 3 immunizations, and the tolerability and efficacy of 3 immunizations are evaluated.

Expansion cohort phase: Based on the safety and efficacy data of the dose escalation phase, combined with safety and immune effect indicators, the dosage and sample size of the expansion cohort study were formulated, their safety and efficacy were evaluated, and the appropriate dose was recommended for subsequent clinical trials.

The sample size of the dose escalation test was planned to be 9~18 cases, and the number of cases in the expansion cohort study was estimated according to the data of the previous dose escalation test.

A total of 3 dose groups were set up for Survivin DC cell injection, which were 1×107 DCs, 2×107 DCs, and 3×107 DCs, and the preparation specification was 6ml. Intradermal administration and intravenous administration are allocated according to a ratio of 1:5, 1ml intradermally and 5ml intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological examination confirming cases of WHO Grade 4 glioblastoma multiforme (GBM) with a new diagnosis.
2. Age between 18 and 70 years, regardless of gender.
3. Karnofsky Performance Status (KPS) score of ≥70 before enrollment.
4. Agreement not to receive any treatment for glioblastoma other than radiotherapy, temozolomide, and PERCELLVAC-Sur immunotherapy during the trial.
5. Positive expression of Survivin in immunohistochemistry testing.
6. Female patients must have a negative pregnancy test, and both male and female participants must agree to non-pharmacological contraceptive measures during the trial (from signing the Informed Consent Form [ICF] to 28 days after the last dose).
7. Laboratory tests with the following criteria: a) White blood cell count ≥ 2.0 × 10^3/mm3 (2.0 × 10^9/L) b) Neutrophil count ≥ 1.5 × 10^3/mm3 (1.5 × 10^9/L) c) Platelet count ≥ 100 × 10^3/mm3 (100 × 10^9/L) d) Hemoglobin ≥ 9.0g/dL (90g/L) e) Serum creatinine ≤ 1.5 × the upper limit of normal (ULN) f) Aspartate transaminase (AST) ≤ 3 × ULN g) Alanine transaminase (ALT) ≤ 3 × ULN h) Total bilirubin ≤ 1.5 × ULN i) Coagulation function: International Normalized Ratio (INR) ≤ 1.5 × ULN; Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN
8. Expected survival period of ≥ 14 weeks. 9) Patients or guardians must sign the Informed Consent Form, demonstrating the ability to read and understand the nature of the experimental study.

Exclusion Criteria:

1. Enhanced MRI within 72 hours after tumor surgery shows residual parts with a diameter exceeding 1cm compared to preoperative remnants.
2. Use of 5-aminolevulinic acid dye during surgery.
3. Failure to complete the prescribed standard 6-week total dose of conformal radiotherapy at 2/3 dose, and cumulative 5 weeks of temozolomide concurrent chemotherapy.
4. Time interval exceeding 50 days from the end of surgery to the start of the 6-week concurrent chemoradiotherapy.
5. Disease progression discovered before the start of treatment after synchronous chemoradiotherapy.
6. Allergic history to the active ingredients or excipients of any investigational drug, including chloride sodium injection containing 10% human serum albumin, penicillin, and ampicillin.
7. Presence of other malignant tumors.
8. Pregnant or lactating women.
9. Corticosteroid (such as dexamethasone) usage exceeding 2mg/day within 30 days before enrollment or during the treatment period, with a single dose interval exceeding 10mg.
10. Need for immunosuppressive agents.
11. Acute infection or unexplained fever: Active viral, bacterial, or fungal infections requiring special treatment (such as antibiotic therapy), or unexplained fever with a temperature exceeding 38℃.
12. Concomitant severe or unstable diseases in the heart, lungs, liver, kidneys, and hematopoietic system. a) Positive for human immunodeficiency virus (HIV), syphilis (spirochete of syphilis), hepatitis A virus (HAV), hepatitis B virus (HBV), or hepatitis C virus (HCV), and HTLV-1/2 (human T-cell leukemia virus), cytomegalovirus (CMV) infections. b) Symptomatic congestive heart failure, unstable angina, arrhythmia. c) Acute myocardial infarction within the last 6 months. d) Presence of severe mental illness or neurological damage, poor patient compliance, or lack of autonomy. e) Neurological diseases, diffuse leptomeningeal diseases, and concomitant neurodegenerative diseases. f) Chronic obstructive pulmonary disease exacerbation requiring hospitalization or other respiratory diseases. g) Immunodeficiency or autoimmune diseases, such as systemic lupus erythematosus, polymyositis, insulin-dependent diabetes, etc.
13. Inability or unwillingness to undergo magnetic resonance imaging (MRI) scans.
14. Participation in any clinical trial within the last 3 months.
15. Investigator's judgment that participation in the clinical trial is not appropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28 days
  The following adverse events that occurred within 28 days after the first dose to the third dose, as judged by the investigator, to be related to the study drug

SECONDARY OUTCOMES:
Progression Free Survival Progression Free Survival | 2 years
  The time from the date of first dose to the occurrence of disease progression or death due to any cause
Overall Survival | 2 years
  The time from the date of first dose to death due to any cause in the subject
Immune effect | 84 days
  Anti-Sauvignon antibody test;
Cytokine | 56 days
  Cytokine (IL-6, IL-8, IL-10, TNF-α, IFN-γ, TGF-β) detection;
Specific T cell responses | 84 days
  Specific T cell responses (Survivin-specific CD4+/CD8+ T cell responses)
DC cell activity and in vivo processes | 35 days
  The quantitative detection of the content of Survivin fusion gene in blood RNA was limited to the quantitative detection of the transcription level of Survivin fusion gene in patients.

IPD SHARING:
Plan to Share IPD: No